CLINICAL TRIAL: NCT05220683
Title: Comparing Two Digital Marking Systems
Brief Title: Digital Marking Systems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VE
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Cataract
Keywords: Astigmatism; Digital Marking Systems
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Verion and Callisto (Experimental): Alignment axis will be analysed with both, the Verion and the Callisto, digital marking system in the same eye of the same patient
  Interventions: Device: digital marking system

INTERVENTIONS:
Device: digital marking system — Verion or Callisto, digital marking system

SUMMARY:
Comparison of the alignment axis of the Alcon Verion and the Zeiss Callisto alignment systems intraoperatively

DETAILED DESCRIPTION:
In most patients undergoing cataract surgery, emmetropia can be achieved by implantation of a monofocal intraocular lens (IOL). However, several studies have shown that approximately 20% to 30% of patients who undergo cataract surgery have a preexisting corneal astigmatism of 1.25 diopters (D) while the prevalence of corneal astigmatism >2.00 D is 8% and over >3.00 D 2.6%. This astigmatism, if not corrected during surgery, leads to postoperative spectacle dependence. In patients without contraindications and a desire to achieve postoperative freedom from spectacles for distance vision, correction of astigmatism can be achieved at the time of surgery by using toric IOLs.

A number of factors relating to corneal astigmatism are critical to lens selection and positioning.The most important factors are the preoperative corneal measurements and the correct alignment of the toric lens itself.

Each degree of deviation results in a 3% reduction in astigmatism correction. The introduction of digital marking systems is intended to minimize the disadvantages of manual marking, such as tilting of the head during marking, incorrect and smudged marking. In addition to several different manual marking methods, there is also a range of digital markers which have been proven to be equal or even better than manual marking. These include among others the Callisto Eye with Z-Align and the Alcon VERION Digital Marker. The principle of these digital marking systems is based on a preoperative photo which is recorded in the course of biometry where the keratometry values are obtained. In the further course, the steep axis is determined on the basis of this image and the target axis is projected on to the eye intraoperatively. Beside the ideal implantation axis for the T-IOL, the size of the capsulorhexis and position, as well as incision placement can be displayed.

In the course of this study, we will investigate the alignment axis of the two most used digital guidance systems from Alcon and Zeiss. A head to head comparison has already been carried out by Hura et al. in 2017.

15 eyes of 15 patients will be included into this study. There will only be one preoperative study visit, on the day of surgery, where reference pictures with a slitlamp camera and the biometers will be taken.

ELIGIBILITY:
Inclusion Criteria:

* age-related cataract and scheduled for cataract surgery
* age 21 or older
* written informed consent prior to surgery

Exclusion Criteria:

* dense cataract or corneal pathology that would significantly influence the measurements
* previous ocular surgery, ocular inflammation, or ocular trauma
* nystagmus or pathologies that might affect patient's fixation
* pregnancy
* corneal astigmatism > 1.5 dpt. or need for a toric IOL

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Alignment axis | 24 months
  Difference in aligment axis will be assessed with the Verion and the Callisto digital marking system

SECONDARY OUTCOMES:
Loss of Tracking | 24 months
  Loss of Tracking will be analysed during the different steps of surgery
Luminance | 24 months
  Luminance necessary for registration will be analysed using a luxmetre

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zeilinger J, Schlatter A, Ruiss M, Bayer N, Kronschlager M, Findl O. Comparison of two digital alignment systems for toric intraocular lens implantation. BMJ Open Ophthalmol. 2024 Sep 16;9(1):e001875. doi: 10.1136/bmjophth-2024-001875. PMID 39284678